CLINICAL TRIAL: NCT01304498
Title: A Randomized, Double-Blinded, Controlled With GARDASIL (Human Papillomavirus Vaccine [Types 6, 11, 16, 18] (Recombinant, Adsorbed)), Phase III Clinical Trial to Study the Immunogenicity and Tolerability of V503 (9-Valent Human Papillomavirus (HPV) Vaccine) in Preadolescent and Adolescent Girls (9- to 15-year-old)
Brief Title: Immunogenicity and Tolerability of V503 Versus GARDASIL (V503-009)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V503-009; GDS01C (Other: MCMVaccBV (SPMSD) Protocol Number); 2010-023393-39 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Human Papillomavirus
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- V503 (Experimental): 9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine, 0.5-mL intramuscular injection in 3 dose regimen at Day 1, Month 2, and Month 6
  Interventions: Biological: V503
- GARDASIL (Active Comparator): Quadrivalent HPV [Types 6, 11, 16, and 18] L1 virus-like particle vaccine, 0.5-mL intramuscular injection in 3 dose regimen at Day 1, Month 2, and Month 6
  Interventions: Biological: GARDASIL

INTERVENTIONS:
Biological: V503 — 9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine
  Other Names: 9vHPV vaccine
  Arms: V503
Biological: GARDASIL — Quadrivalent HPV [Types 6, 11, 16, and 18] L1 virus-like particle vaccine
  Other Names: qHPV vaccine
  Arms: GARDASIL

SUMMARY:
Primary objective:

• To demonstrate that administration of V503 induces non-inferior Geometric Mean Titers (GMTs) (for serum anti-HPV16 and anti-HPV18) compared to GARDASIL.

Secondary objectives:

* To evaluate the tolerability of V503 in 9-15 year-old girls.
* To summarize humoral immune response (anti-HPV 6, 11, 16, 18) induced by V503 or GARDASIL.

ELIGIBILITY:
Inclusion Criteria:

* Female from 9 to 15 years old.
* Good physical health.

Exclusion Criteria:

* Known allergy to any vaccine component.
* History of severe allergic reaction.
* Thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
* Pregnant subject.
* Immunocompromised or immunodeficient subject.
* Splenectomy.
* Receipt of medication / vaccine that may interfere with study assessment.
* Fever
* History of a positive test for HPV, prior receipt of HPV vaccine or prior participation to HPV trial.
* Any condition that might interfere with study assessment.

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2011-02-23 (Actual); Primary Completion 2011-12-20 (Actual); Study Completion 2011-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Vesikari T, Brodszki N, van Damme P, Diez-Domingo J, Icardi G, Petersen LK, Tran C, Thomas S, Luxembourg A, Baudin M. A Randomized, Double-Blind, Phase III Study of the Immunogenicity and Safety of a 9-Valent Human Papillomavirus L1 Virus-Like Particle Vaccine (V503) Versus Gardasil(R) in 9-15-Year-Old Girls. Pediatr Infect Dis J. 2015 Sep;34(9):992-8. doi: 10.1097/INF.0000000000000773. PMID 26090572
- [Derived] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 603 participants were screened and 600 were randomized
Period: Overall Study
Arm/Group | V503 | GARDASIL
Started | 300 | 300
Received ≥1 Dose | 300 | 300
Completed | 294 | 295
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | V503 | GARDASIL | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.6 (1.9) | 12.6 (1.9) | 12.6 (1.9)
Age, Customized [Number; unit: Participants]
  9 to 12 years old | 150 | 150 | 300
  13 to 15 years old | 150 | 150 | 300
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 300 | 600
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) to HPV Types 16 and 18
Description: Serum antibodies to HPV types 16 and 18 were measured with a Competitive Luminex Immunoassay.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: All randomized participants. The n values are participants who received all 3 vaccinations within acceptable day ranges, had Month 7 serology to the HPV type within acceptable day ranges, were seronegative to the HPV type at Day 1, and had no protocol violations that interfered with evaluation of immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 300 | 300
milli Merck Units/mL
  HPV Type 16 (n=276, 270) | 6739.5 [6134.5 to 7404.1] | 6887.4 [6220.8 to 7625.5]
  HPV Type 18 (n=276, 269) | 1956.6 [1737.3 to 2203.7] | 1795.6 [1567.2 to 2057.3]
Statistical Analysis 1: Comparison: V503 vs GARDASIL; HPV Type 16; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.67; p < 0.001, ANOVA; GMT Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11] — GMT ratio = GMT (V503) / GMT (Gardasil)
Statistical Analysis 2: Comparison: V503 vs GARDASIL; HPV Type 18; Test type: Non-Inferiority or Equivalence — Non-inferiority required that the lower bound of the two-sided confidence interval (CI) of the GMT ratio was >0.67; p < 0.001, ANOVA; GMT Ratio = 1.08, 95% CI 2-sided [0.91 to 1.29] — GMT ratio = GMT (V503) / GMT (Gardasil)

2. Secondary Outcome: GMTs to HPV Types 6 and 11
Description: Serum antibodies to HPV types 6 and 11 were measured with a Competitive Luminex Immunoassay.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 300 | 300
milli Merck Units/mL
  HPV Type 6 (n=273, 261) | 1679.4 [1518.9 to 1856.9] | 1565.9 [1412.2 to 1736.3]
  HPV Type 11 (n=273, 261) | 1315.6 [1183.8 to 1462.0] | 1417.3 [1274.2 to 1576.5]

3. Secondary Outcome: Percentage of Participants Who Are Seropositive for HPV Types 6/11/16/18
Description: Serum antibodies to HPV types were measured with a Competitive Luminex Immunoassay. The serostatus cutoffs (milli Merck Units/mL) for HPV types were as follows: HPV Type 6: ≥30; HPV Type 11: ≥16; HPV Type 16: ≥20; HPV Type 18: ≥24. The percentage of participants who were seropositive according to these cutoffs was assessed.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 300 | 300
Percentage of participants
  HPV Type 6 (n=273, 261) | 100 [98.7 to 100] | 100 [98.6 to 100]
  HPV Type 11 (n=273, 261) | 100 [98.7 to 100] | 100 [98.6 to 100]
  HPV Type 16 (n=276, 270) | 100 [98.7 to 100] | 100 [98.6 to 100]
  HPV Type 18 (n=276, 269) | 100 [98.7 to 100] | 100 [98.6 to 100]

4. Secondary Outcome: Percentage of Participants With One or More Adverse Events
Description: An adverse event is defined as any unfavourable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine, is also an adverse event. The percentage of participants with one or more adverse events was assessed.
Time Frame: Up to Month 7
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 299 | 300
Percentage of participants | 96.0 [87.9 to 94.5] | 93.7 [84.1 to 91.7]

5. Secondary Outcome: Percentage of Participants With One or More Injection-site Adverse Reactions
Description: The percentage of participants with one or more injection-site adverse reactions (solicited or unsolicited) was assessed.
Time Frame: Up to 5 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 299 | 300
Percentage of participants | 91.6 [87.9 to 94.5] | 88.3 [84.1 to 91.7]

6. Secondary Outcome: Percentage of Participants With One or More Systemic Adverse Events
Description: The percentage of participants with one or more systemic adverse events was assessed.
Time Frame: Up to 15 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 299 | 300
Percentage of participants | 47.5 [41.7 to 53.3] | 52.0 [46.2 to 57.8]

7. Secondary Outcome: Percentage of Participants With Maximum Oral Temperature ≥37.8°C
Description: The percentage of participants with maximum oral temperature ≥37.8°C was assessed.
Time Frame: Up to 15 days after any vaccination
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 299 | 300
Percentage of participants | 6.7 [4.1 to 10.1] | 3.3 [1.6 to 6.0]

8. Secondary Outcome: Percentage of Participants With One or More Serious Adverse Events
Description: A serious adverse event is an adverse event that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is a cancer, or may jeopardize the participant and may require medical or surgical intervention. The percentage of participants with one or more serious adverse events was assessed.
Time Frame: Up to Month 7
Population: All participants who received at least one study vaccination and had safety follow-up data
Measure: Number; unit: Percentage of participants
Arm/Group | V503 | GARDASIL
Number analyzed (Participants) | 299 | 300
Percentage of participants | 0.3 | 0.7

ADVERSE EVENTS:
Time Frame: All adverse events: up to 15 days after each vaccination; serious adverse events: up to Month 7
Arm/Group | V503 | GARDASIL
Serious Adverse Events (participants affected / at risk) | 1/299 | 2/300
Other Adverse Events (participants affected / at risk) | 280/299 | 274/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V503 (N=299) | GARDASIL (N=300)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V503 (N=299) | GARDASIL (N=300)
Nausea (Gastrointestinal disorders) | 16 (17) | 16 (17)
Injection-site erythema (General disorders) | 102 (132) | 88 (129)
Injection-site pain (General disorders) | 269 (675) | 266 (626)
Injection-site swelling (General disorders) | 144 (226) | 109 (160)
Pyrexia (General disorders) | 22 (23) | 17 (17)
Nasopharyngitis (Infections and infestations) | 5 (7) | 16 (18)
Headache (Nervous system disorders) | 57 (84) | 57 (93)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.